CLINICAL TRIAL: NCT06147518
Title: An Open Label Randomized Control Trial to Compare the Safety and Efficacy of Dapagliflozin Plus Metformin Versus Sitagliptin Plus Metformin for Treatment of Diabetes in Patients With Compensated and Stable Decompensated Cirrhosis
Brief Title: To Compare the Safety and Efficacy of Dapagliflozin Plus Metformin Versus Sitagliptin Plus Metformin for Treatment of Diabetes in Patients With Compensated and Stable Decompensated Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-68
Record Dates: First submitted 2023-11-16; First posted 2023-11-27 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Compensated Cirrhosis; Decompensated Cirrhosis
MeSH Terms: interventions — Metformin; Sitagliptin Phosphate; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin with Sitagliptin (Active Comparator): Metformin: 1.5g/d CTPA,1g/d CTPB Sitagliptin: Assess HbA1c/HBSG at 8 weeks, increase sitagliptin to 100 mg if HbA1c>7%
  Interventions: Drug: Metformin; Drug: Sitagliptin
- Metformin with Dapagliflozin (Experimental): Metformin: 1.5g/d CTPA,1g/d CTPB
  Dapagliflozin: Assess HbA1c/HBSG at 8 weeks, increase dapagliflozin to 10 mg if HbA1c>7%
  Interventions: Drug: Metformin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Metformin — Metformin: 1.5g/d CTPA,1g/d CTPB
Drug: Sitagliptin — Sitagliptin: Assess HbA1c/HBSG at 8 weeks, increase sitagliptin to 100 mg if HbA1c>7%
  Arms: Metformin with Sitagliptin
Drug: Dapagliflozin — Assess HbA1c/HBSG at 8 weeks, increase Dapagliflozin to 10 mg if HbA1c>7%
  Arms: Metformin with Dapagliflozin

SUMMARY:
Diabetes prevalence is increasing among cirrhotics and use of OAD in cirrhotics is limited because of risk of hypoglycaemia and other adverse effects, therefore in this study we would be using OAD in the form of Sitagliptin or Dapagliflozin to look for glycemic response as well as to look for other benefits such as weight reduction and improvement in lipid parameters.

DETAILED DESCRIPTION:
Hypothesis In patients with cirrhosis and T2DM with poor glycemic control on metformin requiring dual therapy, Dapagliflozin is safe and superior to Sitagliptin in achieving glycemic control. Moreover, Dapagliflozin use leads to improvement in parameters of metabolic dysfunction, clinical decompensation and cardio-renal protection.

Aim compare the safety and efficacy of metformin plus sitagliptin compared to metformin plus dapagliflozin in effective glycemic control and improvement in parameters of metabolic dysfunction, cirrhosis complications and organ dysfunction at 24 weeks.

Study population:Patients with compensated and stable decompensated cirrhosis and age 18-70 years with CTP 5-8

Study design: A prospective, randomized, single center open label study

The study will be conducted on the consecutive patients with liver cirrhosis and type 2 diabetes mellitus seen at the outpatient clinics of Department of Hepatology, ILBS

Sample size: 200 Assuming that 40% people had HbA1c <7 in Dapagliflozin and 25% in sitagliptin.Alpha = 5%,Power = 80%,Need to enroll total 200 cases(100 in each arm), Drop rate = 10%,Total enrollment = 100 cases (80 each arm).

Randomization by block randomization method taking block size as 10 Intervention: This RCT will be conducted at ILBS New Delhi

Monitoring and assessment: Monitoring will be done for all the parameters of the objective. Documentation will be done for any adverse effects which will happen.

Adverse effects: to be monitored

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Child A/B Liver cirrhosis in outpatient setting
3. T2DM patients who have not used any glucose-lowering agents within 8 weeks before consenting, or those who have only used metformin, in addition to diet and exercise
4. HbA1c level of 7.1% or higher but no more than 9.0%
5. BMI of 23 kg/m2 or higher
6. patients who can be monitored closely for medication compliance
7. patients who provide written informed consent.

Exclusion Criteria:

1. Age <18 years
2. Post renal or liver transplantation
3. CTP C / ACLF
4. Intrinsic/structural kidney disease, obstructive uropathy, ADPKD, Anatomic urologic defects that predispose to urinary tract infection
5. Active sepsis / SBP at enrollment
6. Grade II/III/IV HE
7. Pregnancy or Lactating mother
8. Known CKD, obstructive uropathy
9. Patient on MV, NIV, systemic sepsis and shock
10. Lack of informed consent
11. Prior intolerance or S/E to SGLT-2i or DPP4i
12. patients with type 1 diabetes or secondary diabetes
13. patients with medical history of diabetic ketoacidosis
14. patients with medical history of myocardial infarction, cerebral infarction, or stroke within 12 weeks before consent to the study
15. estimated glomerular filtration rate (eGFR) less than 45 mL/min/1.73 m2
16. unstable hypertension or dyslipidemia within 12 weeks before consent to the study
17. HB <9 g/L, patients with haemoglobinopathy, acute hemolysisStudy period: one year after ethical approval.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with glycemic control at 24 weeks (HBA1c <7.0 %) | 24 weeks

SECONDARY OUTCOMES:
Percentage of patients with glycemic control at 8 and 16 weeks (HBA1c <7.0 %) | 8 and 16 weeks
Ideal body weight loss of ≥3% relative to baseline at 24 week | 24 weeks
Incidence and frequency of hypoglycemia (BS <54 mg/dl) episodes | 8 weeks
Incidence and frequency of hypoglycemia (BS <54 mg/dl) episodes | 16 weeks
Incidence and frequency of hypoglycemia (BS <54 mg/dl) episodes | 24 weeks
Changes in HbA1c at 24 week relative to baseline | 24 weeks
Changes in BMI at 24 week relative to baseline | 24 weeks
changes in Blood insulin at 24 week | 24 weeks
changes in lipid profile at 24 week | 24 weeks
Change in ALT at 8, 16 and 24 week | 8, 16 and 24 week
Change in HVPG at 24 week compared to baseline | 24 weeks
Change in LSM at 24 week compared to baseline | 24 weeks
Change in SSM at 24 week compared to baseline | 24 weeks
Incidence of urinary protein excretion at 8, 16 and 24 weeks | 8, 16 and 24 weeks
Incidence of serum creatinine at 8, 16 and 24 weeks | 8, 16 and 24 weeks
Number of patients with Complications of cirrhosis (ascites, HE, Bleed, AKI, Infection) at 24 week | 24 weeks
Medicine adherence rate in both groups | 24 weeks
Adverse effects to study drugs in both groups | 24 weeks
Number of patients with Mortality/ Liver transplantation in both groups | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Rakesh Kumar Jagdish, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided